CLINICAL TRIAL: NCT04753138
Title: The Outcome of Non-surgical Root Canal Treatment Using Sealer-based Obturation With Calcium Silicate Sealer vs. Warm Vertical Compaction With AH+ Sealer. A Randomized Controlled Clinical Trial
Brief Title: Outcome of SBO With Calcium Silicate Sealer vs WVC With Resin Based Sealer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait Institute for Medical Specialization (Other Government)
Collaborators: Ministry of Health, Kuwait (Other Government); Kuwait Foundation for the Advancement of Sciences (Unknown)
Responsible Party: Principal Investigator, Fahad Alzoubi, Chair of Faculty of Dentistry, Kuwait Institute for Medical Specialization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fahadmz
Record Dates: First submitted 2021-01-26; First posted 2021-02-15 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Root Canal Obturation; Root Canal Filling; Sealer-based Obturation; Randomized Clinical Trial; Postoperative Pain; Resin Based Sealer; Warm Vertical Compaction
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Permuted block randomization (of block size = only known to statistician) will be used to randomly select 212 subjects (106 subjects in each group). Statistical software (NCSS, LLC© ver. 2020) will be utilized to generate the randomization list and subjects will be assigned to the selected treatment group accordingly.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the type of treatment they receive to reduce bias in the reporting of postoperative pain.
  Since it is not possible to blind the care providers, they will only be informed of the type of treatment once full chemo-mechanical debridement has been completed and the tooth is ready to be obturated. This would reduce care provider bias.
  Assessors will be blinded to the treatment option to reduce bias during the assessment of healing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBO with calcium silicate sealer (Experimental): The teeth will be obturated with the single cone technique and BC sealer
  Interventions: Device: TotalFill Bioceramic Sealer
- WVC with resin based sealer (Active Comparator): The teeth will be obturated with warm vertical compaction and AH+ sealer
  Interventions: Device: AH+ Sealer

INTERVENTIONS:
Device: TotalFill Bioceramic Sealer — It will be used in conjunction with TotalFill® bioceramic impregnated gutta percha points for the obturation of root canals. It is dispensed through a fine disposable syringe into the root canals during obturation.
  Arms: SBO with calcium silicate sealer
Device: AH+ Sealer — It consists of 2 pastes that are mixed together in equal amounts before it is used in conjunction with gutta percha points for obturation during root canal treatment.
  Arms: WVC with resin based sealer

SUMMARY:
A single blinded randomized controlled trial. 212 subjects (teeth), 106 in each of the 2 groups will be recruited from the patients referred to Kuwait Board of Endodontics for primary root canal treatment. The aim is to compare the outcome of sealer-based obturation (SBO) with calcium silicate sealer versus warm vertical compaction (WVC) and resin based sealer.

Preoperative PA radiograph and CBCT will be taken. A 1 year follow up period will be arranged and another PA radiograph and CBCT will be taken. The preoperative, postoperative and review clinical and radiographic data will be analyzed

DETAILED DESCRIPTION:
Aims and Objectives

* To compare the clinical outcome of the SBO with WVC in non-surgical root canal treatment.
* To compare the radiographic outcome of the SBO with WVC in non-surgical root canal treatment using periapical radiographs and CBCT scans.
* To assess the difference in postoperative pain between the 2 groups.
* To assess the difference in the time required to complete the obturation between the 2 groups.

Materials and Methods

* Patients who are referred to the Kuwait Board of Endodontics for non-surgical root canal treatment and fulfil the inclusion/exclusion criteria of the study will be included
* Pre-operative periapical radiograph, CBCT scan and 11-point Numerical Rating Scale (NRS) will be taken.
* Upon completion of root canal instrumentation, the participants will be randomly allocated to either Group A: obturation using SCCS or Group B: obturation using WVC. The participants will be blinded to the type of treatment received and the clinician will only be informed of the obturation method once the canal/canals are ready for obturation.
* All teeth will then be restored definitively.
* The participants will be contacted via telephone 1, 3 and 7 days post-treatment to report their NRS pain score.
* The participants will be recalled after 1 year for clinical and radiographic assessment using periapical radiograph and CBCT scan.
* The participants will then be followed-up annually for up to 4 years.
* Statistical analysis will be performed.
* The design of the study will conform to the CONSORT statement.

Statistical and Analytical Plans

Sample size estimation for the treatment outcome was performed using PASS 2019 computer software, utilizing information from previous studies on healing outcome after initial endodontic therapy. For a two independent-samples t-test of proportions, at power of 80% and 5% significance level for two-tailed test, detecting a 10% difference of healing rate required a sample size of 148 teeth. Adjusting for a dropout rate of 30%, the required sample size was 212 teeth. The slightly high 30% dropout rate is anticipated because most of the patients we treat are non-Kuwaiti nationals and their presence in the country after 1 year is not guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a classification of I or II on the American Society of Anesthesiologists (ASA) physical status classification system
* Participants must not have known allergies to any materials used in the study
* Participants must agree to participate in the study by signing a consent form
* All types of permanent teeth are included (incisors, canines, premolars & molars)
* The teeth must be restorable and have fully formed roots with no advanced periodontal disease
* In the event that a patient has more than 1 tooth eligible for the study, only one tooth on the left and/or right side of the mouth will be selected at random. A maximum of 2 teeth per participant can be included in the study

Exclusion Criteria:

* ASA classification of III or more
* Pregnant women
* Advanced periodontal disease or teeth with more than 5mm probing
* Teeth with incomplete root formation or root resorption
* Teeth with adjacent teeth that require RCT
* Previously root canal treated teeth
* Teeth with a history of trauma
* Teeth that have poor restorative prognosis
* Teeth requiring extensive prosthodontic rehabilitation
* Cracked teeth

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Assessment of radiographic healing with periapical (PA) radiographs using Orstavik's PAI | Comparison of of periapical lesion size at baseline and 12 months
  Proportion t-test will be carried to compare the proportion of study subjects with improved apical lesion size between the two treatment groups. Odds ratio with 95% confidence interval will be reported. Logistic regression analysis adjusted for the stratification variables (gender) and other confounding factors (namely patency, extrusion of sealer or GP, short fill, voids, pre-op apical size, pre-op clinical symptoms and number of C&S visits). Orstavik's periapical index (PAI) will be used as the outcome measure
Assessment of radiographic healing with Cone beam computed tomography (CBCT) scans using Estrela's PAI based on CBCT | Comparison of of periapical lesion size at baseline and 12 months
  Proportion t-test will be carried to compare the proportion of study subjects with improved apical lesion size between the two treatment groups. Odds ratio with 95% confidence interval will be reported. Logistic regression analysis adjusted for the stratification variables (gender) and other confounding factors (namely patency, extrusion of sealer or GP, short fill, voids, pre-op apical size, pre-op clinical symptoms and number of C&S visits). Estrela's (periapical index) PAI based on CBCT will be used as outcome measure
Assessment of clinical outcome by assessing the resolution/persistence/development of clinical signs and symptoms | Comparison at baseline and 12 months
  The examiner will label the teeth as having a normal clinical outcome (absence of pain, swelling and other symptoms, no sinus tract, no loss of function) or showing signs and symptoms clinical outcome (The tooth is associated with signs and/or symptoms of infection)

SECONDARY OUTCOMES:
Comparison of the postoperative pain score | 1, 3 and 7 days postoperatively
  11 point Numerical Rating Scale (NRS) will be used. The participants will be given an NRS sheet to complete. They will be asked to choose a number between 0 'No Pain' and 10 'Worst imaginable pain' that best represents your pain intensity.
Comparison of the time required to complete obturation between the 2 groups | Intra-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alzoubi, M.Endo, Principal Investigator — Kuwait Board of Endodontics
Locations (1):
- Specialized Dental Center, Kuwait City, Kuwait

REFERENCES:
- [Derived] Alzoubi F, Alajmi S, Alkandari A, Alqahtani S, Alanezi A, Setzer FC. Post-operative pain in non-surgical root canal treatment after sealer-based obturation versus warm vertical compaction: A randomized clinical trial. Int Endod J. 2024 Sep;57(9):1168-1179. doi: 10.1111/iej.14102. Epub 2024 May 30. PMID 38813933